CLINICAL TRIAL: NCT03278379
Title: A Phase II Study of Avelumab in Unresectable/Metastatic, Progressive Grade 2-3 Neuroendocrine Tumors
Brief Title: Avelumab in G2-3 NET
Acronym: NET-002
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 414-2016
Record Dates: First submitted 2017-08-23; First posted 2017-09-11 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-11

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intervention Arm (Experimental): Treatment with Avelumab
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Avelumab — Avelumab will be administered intravenously as an infusion, at a dose of 10 milligram per kilogram once every 2 weeks, until occurence of progressive disease, unacceptable toxicity, or any of the other criteria for withdrawal listed in the protocol .

SUMMARY:
This is a single-center, single-arm, open-label, phase II trial to evaluate the efficacy and safety of avelumab in subjects with unresectable or metastatic, Grade 2-3, well-differentiated neuroendocrine.tumour.

ELIGIBILITY:
Inclusion Criteria:

* Adults (males or females), aged 18 years or older with pathologically confirmed, advanced (unresectable or metastatic) neuroendocrine tumour from a gastroenteropancreatic or lung source. Both participants with functional NETs and those with nonfunctional NETs shall be eligible for this study.
* Histologically confirmed, WHO Grade 2-3, well-differentiated NETs of gastroenteropancreatic or lung origin.
* Has received 0,1 or 2 prior lines of systemic therapy (chemotherapy, PRRT, targeted therapies such as everolimus or sunitinib). Somatostatin analogues are not considered a line of therapy for the purposes of this criterion.
* Radiological documentation of disease progression within 24 weeks of study enrolment. Disease progression must be demonstrated on two scans less than one year apart.

  * Participants previously treated with any systemic therapies are eligible to enroll if disease progression is documented during or after their last treatment.
* Measurable disease as assessed by CT scan of the chest, abdomen and pelvis which is suitable for accurate repeated measurements (according to RECIST v1.1).
* ECOG performance status 0-2.
* Adequate bone marrow function (ANC > 1.5 x 109/L; Platelets >100 x109/L; haemoglobin > 90 g9/L).
* Adequate liver function defined by a total bilirubin level ≤1.5xULN and AST and ALT levels ≤2.5xULN for participants (or AST and ALT levels ≤ 5xULN for participants with documented metastatic disease to the liver).
* Adequate renal function defined by an estimated creatinine clearance ≥ 30 mL/min according to the Cockcroft-Gault formula (or local institutional standard method).
* Willing and able to comply with all study requirements, including timing and/or nature of treatment and required assessments.
* Signed, written informed consent.
* Evidence of post-menopausal status, or negative urine or serum pregnancy test for female pre-menopausal participants (within approximately 14 days prior to enrolment). Women will be considered post-menopausal if they have been amenorrhoeic for 12 months without an alternative medical explanation.
* Highly effective contraception for both male and female participants if the risk of conception exists (note: The effects of the IP on the developing human fetus are unknown; thus, women of childbearing potential and men able to father a child must agree to use 2 highly effective contraceptions, defined as methods with a failure rate of less than 1% per year. Highly effective contraception is required at least 28 days prior, throughout and for at least 60 days after avelumab treatment.)

Exclusion Criteria:

* Grade 1 NET or Grade 3 poorly-differentiated neuroendocrine carcinoma, or mixed adenoneuroendocrine carcinomas (MANEC)
* NETs confirmed to be from primaries other than the gastrointestinal tract, pancreas, or lung
* Prior use of PD-1, PD-L1 or CTLA-4 inhibitors
* Life expectancy of ≤3 months
* Concurrent treatment with other anticancer therapy (except somatostatin analogues for the purposes of functional control). Participants on somatostatin analogues for anti-proliferative therapy should have this therapy ceased, and would be eligible for enrolment if they have not received somatostatin analogues in the past 14 days.
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent, with exception to:
* Subjects with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible
* Active infection requiring systemic therapy.
* History of primary autoimmunodeficiency
* Current use of immunosuppressive medication, EXCEPT for the following: a. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); b. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; c. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
* Prior organ transplantation, including allogeneic stem cell transplantation
* Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
* Major surgery in the 2 weeks prior to randomization. Surgery with intent to debulk metastatic disease is allowed, as long as there is sufficient residual disease for RECIST measurements (see inclusion criteria 5).
* Participants with prior or concurrent malignancy except for the following: adequately treated basal cell or squamous cell skin cancer, or other adequately treated in situ cancer, or any other cancer from which the patient has been disease free for three years.
* All participants with brain metastases and any of the following:

  * They have not received local treatment to known brain metastases
  * They have been clinically unstable in the 2 weeks prior to enrolment
  * Requirement for treatment with systemic steroids exceeding the equivalent of 10mg oral prednisone per day
  * Ongoing neurological symptoms related to brain metastases
  * Leptomeningeal metastases
* Pregnancy, lactation, or inadequate contraception.
* Significant acute or chronic infections including, among others:

  * Known history of positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
  * Positive test for HBV surface antigen and / or confirmatory HCV RNA (if anti-HCV antibody tested positive)
  * Active tuberculosis
  * Testing for these diseases is not mandatory unless clinically indicated.
* Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v4.03 Grade ≥ 3)
* Persisting toxicity related to prior therapy of Grade >1 NCI-CTCAE v 4.03; however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable.
* Known alcohol or drug abuse
* Other severe acute or chronic medical conditions including colitis, inflammatory bowel disease, pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
* Any psychiatric condition that would prohibit the understanding or rendering of informed consent
* Vaccination within 4 weeks of the first dose of avelumab and while on trial, except for administration of inactivated vaccines
* Inability to obtain sufficient tumour tissue (whether archival or fresh) for PD-L1 testing. A core biopsy, endoscopic biopsy or surgical resection specimen shall be considered adequate tissue; a fine needle aspirate/biopsy will be considered insufficient tissue.
* Prior treatment for study indication with:

  * Peptide Receptor Radiouclide Therapy (PRRT) administered within 3 months of enrolment
  * Hepatic intra-arterial embolization, radio-frequency ablation, or cryoablation within 4 weeks of enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to 2 years
  The overall response rate will be defined as the number of participants with confirmed complete response or partial response (CR or PR) recorded as the best response over the study period, divided by the number of participants evaluable for response as defined by RECIST version 1.1.

SECONDARY OUTCOMES:
Disease control rate (DCR) | Up to 2 years
  The DCR will be defined as the number of patients with confirmed CR, PR or stable disease (SD) recorded as the best response over the study period, divided by the number of participants evaluable for response as defined by RECIST version 1.1.
Duration of response | Up to 2 years
  Time from documentation of tumour response to disease progression
Progression-free survival (PFS) | Up to 2 years
  PFS is defined as the time from first administration of study drug to the date of documented confirmed progression or death, whichever comes first
Overall survival (OS) | Up to 2 years
  OS is defined as the time from first administration of drug to date of death.
Rates of treatment-emergent adverse events as defined by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.03 | Up to 90 days after the last dose is administered
ORR by irRECIST version 1.1 | Up to 2 years
DCR by irRECIST version 1.1 | Up to 2 years
Duration of response by irRECIST version 1.1 | Up to 2 years
PFS by irRECIST version 1.1 | Up to 2 years
OS at 1 year | 1 year
OS at 2 years | 2 years
PFS at 1 year | 1 year
PFS at 2 years | 2 years

OTHER OUTCOMES:
Correlation of PD-L1 status with response to avelumab | Up to 2 years
Correlation of mutational load and T-cell repertoire analysis with response to avelumab | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Simron Singh, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Chan DL, Rodriguez-Freixinos V, Doherty M, Wasson K, Iscoe N, Raskin W, Hallet J, Myrehaug S, Law C, Thawer A, Nguyen K, Singh S. Avelumab in unresectable/metastatic, progressive, grade 2-3 neuroendocrine neoplasms (NENs): Combined results from NET-001 and NET-002 trials. Eur J Cancer. 2022 Jul;169:74-81. doi: 10.1016/j.ejca.2022.03.029. Epub 2022 May 2. PMID 35504244